CLINICAL TRIAL: NCT01102764
Title: Prolonged Exposure (PE) for PTSD: Telemedicine vs. In Person
Brief Title: Prolonged Exposure (PE) for Post Traumatic Stress Disorder (PTSD): Telemedicine Versus In Person
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Pennsylvania (Other); University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IAC 09-040; 19695 (Other: Medical University of South Carolina IRB)
Record Dates: First submitted 2010-03-17; First posted 2010-04-13 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2018-11

CONDITIONS: PTSD
Keywords: Anxiety Disorders: PTSD; Prolong Exposure (PE); Telemedicine; cost effectiveness; deployment related problems; mental health care delivery
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: PE via telemedicine (Experimental): PE via telemedicine
  Interventions: Behavioral: Telemedicine
- Arm 2: PE in person (Active Comparator): PE in person
  Interventions: Behavioral: In Person

INTERVENTIONS:
Behavioral: Telemedicine — Prolonged Exposure (PE) therapy provided at patients house via telemedicine
  Arms: Arm 1: PE via telemedicine
Behavioral: In Person — PE therapy delivered in person at the VAMC
  Arms: Arm 2: PE in person

SUMMARY:
The present proposal is to study whether Prolonged Exposure (PE) delivered via Telemedicine is as effective as PE delivered In Person for Operation Iraqi Freedom (OIF), Operation Enduring Freedom (OEF) Veterans and Veterans of all theatres, particularly Vietnam era with Post-Traumatic Stress Disorder (PTSD). ).

DETAILED DESCRIPTION:
Project Background/Rationale: Approximately 15 to 17% of current Iraq war Veterans meet full diagnostic criteria for MH problems such as post-traumatic stress disorder (PTSD) (Hoge et al., 2004). Prolonged Exposure (PE) is an empirically supported treatment for PTSD (Foa 1997; Schnurr et al., 2007), and has been adopted by the Department of Veterans Affairs (DOVA) as one of the treatments of choice for the disorder, as evident by the DOVA-sponsored national training of clinicians to use PE. It is therefore important to employ treatment delivery methods that maximize the likelihood that all Veterans in need, including Veterans residing in rural settings, and Veterans who avoid DOVA settings due to the stigma of receiving mental health treatment, will receive interventions such as PE. The May, 2005 Committee on Veterans Affairs, Subcommittee on Health has identified Telemedicine as a DOVA priority area to address this need. The present proposal is to study whether PE delivered via Telemedicine is as effective as PE delivered In Person. Telemedicine has been chosen for its ability to overcome what appear to be two major barriers to mental health care (Frueh et al., 2000): the difficulty that rural-residing Veterans face in reaching VAMC facilities, and the stigma Veterans perceive related to receiving mental health treatment. Indeed, if effective, PE delivered via telemedicine may address the problem inherent in the finding that 42% of those screening positive for PTSD indicate that they are interested in receiving help, but only 25% actually receive services (Hoge, et al., 2006).

Project Objectives: Although effective treatments for PTSD exist and have been adopted by the Veterans Affairs Medical Centers (VAMC), barriers to care of a social (e.g., stigma) and geographic (e.g., rural) nature prevent many Veterans in need from receiving care. Telemedicine might address this need. The major objective of this study is to determine if PE delivered via Telemedicine is as effective as In Person PE in terms of (1) clinical; (2) process; and (3) economic outcomes.

Project Methods: The investigators propose to use a randomized between groups repeated measures (baseline, post-treatment, 3& 6-month followups) design with 226 OIF-OEF Veterans diagnosed with PTSD to assess the relative effectiveness, measured in terms of symptoms, patient satisfaction, and costs, of PE delivered via Telemedicine vs. In Person formats. The investigators hypothesize that no differences (i.e., non-inferiority) between the two formats will be evident in terms treatment gains, patient satisfaction, treatment attrition, patient satisfaction and direct health care costs.

Anticipated Impacts on Veterans Health care: This study will provide important information regarding whether PE delivered via home-based Telemedicine equipment is as effective as traditional In Person delivery of PE for post-traumatic stress disorder. If shown to be as effective as In Person treatment, a new, innovative, and cost effective intervention delivery system for PTSD will have initial empirical support.

ELIGIBILITY:
Inclusion Criteria:

Participants will be 226 male and female:

* Operation Iraqi Freedom, Operation Enduring Freedom (OIF OEF) Veterans, and Veterans of all theatres, particularly Vietnam era Veterans.
* age 21 and above, and
* diagnosed via structured clinical interview with PTSD

Exclusion Criteria:

* Actively psychotic or demented persons,
* individuals with both suicidal ideation and clear intent, and
* individuals meeting full criteria for substance dependence will be excluded from participation

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-10; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron E. Acierno, PhD MS BA, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

REFERENCES:
- [Background] Strachan M, Gros DF, Yuen E, Ruggiero KJ, Foa EB, Acierno R. Home-based telehealth to deliver evidence-based psychotherapy in veterans with PTSD. Contemp Clin Trials. 2012 Mar;33(2):402-9. doi: 10.1016/j.cct.2011.11.007. Epub 2011 Nov 11. PMID 22101225
- [Background] Gros DF, Price M, Strachan M, Yuen EK, Milanak ME, Acierno R. Behavioral activation and therapeutic exposure: an investigation of relative symptom changes in PTSD and depression during the course of integrated behavioral activation, situational exposure, and imaginal exposure techniques. Behav Modif. 2012 Jul;36(4):580-99. doi: 10.1177/0145445512448097. Epub 2012 Jun 7. PMID 22679240
- [Background] Tuerk PW, Wangelin B, Rauch SA, Dismuke CE, Yoder M, Myrick H, Eftekhari A, Acierno R. Health service utilization before and after evidence-based treatment for PTSD. Psychol Serv. 2013 Nov;10(4):401-9. doi: 10.1037/a0030549. Epub 2012 Nov 12. PMID 23148769
- [Background] Price M, Gros DF, Strachan M, Ruggiero KJ, Acierno R. The Role of Social Support in Exposure Therapy for Operation Iraqi Freedom/Operation Enduring Freedom Veterans: A Preliminary Investigation. Psychol Trauma. 2013 Jan 1;5(1):93-100. doi: 10.1037/a0026244. PMID 23869250
- [Background] Gros DF, Gros K, Acierno R, Frueh BC, Moreland L. Relation between treatment satisfaction and treatment outcome in veterans with posttraumatic stress disorder. Journal of psychopathology and behavioral assessment. 2013 Jun 28; 35(4):522-30.
- [Background] Acierno R, Gros DF, Morland L, Greene C, Strachan MK, Egede LE, Tuerk PW, Frueh BC, Myrick H. Delivery of evidence-based psychotherapy via video telehealth. Journal of psychopathology and behavioral assessment. 2013 Dec 1; 35(4):506-521.
- [Background] Gros DF, Price M, Yuen EK, Acierno R. Predictors of completion of exposure therapy in OEF/OIF veterans with posttraumatic stress disorder. Depress Anxiety. 2013 Nov;30(11):1107-13. doi: 10.1002/da.22207. Epub 2013 Oct 21. PMID 24151141
- [Background] Soltis K, Acierno R, Gros DF, Yoder M, Tuerk PW. Post-traumatic stress disorder: ethical and legal relevance to the criminal justice system. J Law Med Ethics. 2014 Summer;42(2):147-54. doi: 10.1111/jlme.12130. PMID 25040378
- [Background] Paul LA, Gros DF, Strachan M, Worsham G, Foa EB, Acierno R. Prolonged Exposure for Guilt and Shame in a Veteran of Operation Iraqi Freedom. Am J Psychother. 2014 Sep 1;68(3):277-286. doi: 10.1176/appi.psychotherapy.2014.68.3.277. PMID 25505798
- [Background] Hernandez-Tejada MA, Zoller JS, Ruggiero KJ, Kazley AS, Acierno R. Early treatment withdrawal from evidence-based psychotherapy for PTSD: telemedicine and in-person parameters. Int J Psychiatry Med. 2014;48(1):33-55. doi: 10.2190/PM.48.1.d. PMID 25354925
- [Background] Yuen EK, Gros DF, Price M, Zeigler S, Tuerk PW, Foa EB, Acierno R. Randomized Controlled Trial of Home-Based Telehealth Versus In-Person Prolonged Exposure for Combat-Related PTSD in Veterans: Preliminary Results. J Clin Psychol. 2015 Jun;71(6):500-12. doi: 10.1002/jclp.22168. Epub 2015 Mar 25. PMID 25809565
- [Background] Badour CL, Gros DF, Szafranski DD, Acierno R. Problems in sexual functioning among male OEF/OIF veterans seeking treatment for posttraumatic stress. Compr Psychiatry. 2015 Apr;58:74-81. doi: 10.1016/j.comppsych.2014.12.012. Epub 2014 Dec 30. PMID 25596624
- [Background] Zhang J, Sheerin C, Mandel H, Banducci AN, Myrick H, Acierno R, Amstadter AB, Wang Z. Variation in SLC1A1 is related to combat-related posttraumatic stress disorder. J Anxiety Disord. 2014 Dec;28(8):902-7. doi: 10.1016/j.janxdis.2014.09.013. Epub 2014 Oct 5. PMID 25445080
- [Background] Pelton D, Wangelin B, Tuerk P. Utilizing Telehealth to Support Treatment of Acute Stress Disorder in a Theater of War: Prolonged Exposure via Clinical Videoconferencing. Telemed J E Health. 2015 May;21(5):382-7. doi: 10.1089/tmj.2014.0111. Epub 2015 Mar 12. PMID 25764266
- [Background] Tuerk PW. Starting from something: augmenting exposure therapy and methods of inquiry. Am J Psychiatry. 2014 Oct;171(10):1034-7. doi: 10.1176/appi.ajp.2014.14070880. No abstract available. PMID 25272341
- [Result] Hershenberg R, Paulson D, Gros DF, Acierno R. Does Amount and Type of Activity Matter in Behavioral Activation? A Preliminary Investigation of the Relationship between Pleasant, Functional, and Social Activities and Outcome. Behav Cogn Psychother. 2015 Jul;43(4):396-411. doi: 10.1017/S1352465813001185. Epub 2014 Mar 13. PMID 24621452
- [Result] Price M, Kuhn E, Hoffman JE, Ruzek J, Acierno R. Comparison of the PTSD Checklist (PCL) Administered via a Mobile Device Relative to a Paper Form. J Trauma Stress. 2015 Oct;28(5):480-3. doi: 10.1002/jts.22037. Epub 2015 Sep 16. PMID 26375277
- [Result] Acierno R, Gros DF, Ruggiero KJ, Hernandez-Tejada BM, Knapp RG, Lejuez CW, Muzzy W, Frueh CB, Egede LE, Tuerk PW. BEHAVIORAL ACTIVATION AND THERAPEUTIC EXPOSURE FOR POSTTRAUMATIC STRESS DISORDER: A NONINFERIORITY TRIAL OF TREATMENT DELIVERED IN PERSON VERSUS HOME-BASED TELEHEALTH. Depress Anxiety. 2016 May;33(5):415-23. doi: 10.1002/da.22476. Epub 2016 Feb 10. PMID 26864655
- [Result] Korte KJ, Allan NP, Gros DF, Acierno R. Differential treatment response trajectories in individuals with subclinical and clinical PTSD. J Anxiety Disord. 2016 Mar;38:95-101. doi: 10.1016/j.janxdis.2016.01.006. Epub 2016 Jan 21. PMID 26874291
- [Result] Acierno RE. Symptoms of posttraumatic stress disorder and major depressive disorder in veterans of Operations Enduring/Iraqi Freedom in comparison with those veterans of other conflicts. Military Behavioral Health. 2016 Apr 25; 4(4):383-389.
- See also: Click here for more information about this study: Prolonged Exposure (PE) for PTSD: Telemedicine vs. In Person — http://www.ptsd.va.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The research team mailed invitation to participate brochures to a VAMC roster of Veterans of all theatres. IRB-approved recruitment flyers were placed throughout the main hospital and surrounding VA clinics. Furthermore, the team accepted direct referrals from VA providers and the Post Traumatic Stress Disorder Clinical Team (PCT).
Pre-assignment Details: There were 150 participants enrolled in the study, and 132 completed at least one session and were thus analyzed. The numbers here reflect those participants who were analyzed because they completed at least 1 treatment session.
Period: Overall Study
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person
Started | 64 | 68
Completed | 43 | 55
Not Completed | 21 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person | Total
Number analyzed (Participants) | 64 | 68 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (14.9) | 42.9 (14.1) | 41.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 63 | 64 | 127
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 23 | 44
  White | 39 | 41 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 64 | 68 | 132
Mean Service Connection Rating [Mean (Standard Deviation); unit: units on a scale] — Veterans can have anywhere from 0% to 100% service connection rating aka "disability compensation." Disability compensation is a monetary benefit paid to Veterans who are determined by VA to be disabled by an injury or illness that was incurred or aggravated during active military service. These disabilities are considered to be service connected. To be eligible for compensation, the Veteran must have been separated or discharged under conditions other than dishonorable.
  units on a scale | 55.8 (35.7) | 51.4 (40.2) | 53.5 (37.9)
Marital Status [Number; unit: participants]
  Never Married | 15 | 15 | 30
  Married | 36 | 37 | 73
  Separated/Divorced | 11 | 12 | 23
  Widowed | 1 | 2 | 3
  Unknown | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Treatment Completion
Description: The major objective of this study is to determine if PE delivered via Telemedicine is as effective as In Person PE in terms of (1) clinical (PTSD and Depression); (2) process (Treatment Satisfaction and Attrition); and (3) economic (Cost) outcomes. Per protocol, participants could have as many as 12 treatment sessions. Per protocol treatment completers completed at least 6 90-minute sessions of Prolonged Exposure either In Person or via Telemedicine. Treatment dropout is defined as initiating treatment but completing fewer than 6 sessions.
Time Frame: 13 weeks
Population: There were 150 participants enrolled in the study, and 132 completed at least one session and were thus analyzed. The numbers here reflect those participants who completed at least one session.
Measure: Mean (Full Range); unit: sessions
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person
Number analyzed (Participants) | 64 | 68
sessions
  Overall Average Number of Sessions Completed | 7.6 [1 to 12] | 8.6 [1 to 12]
  Average Number of Sessions Prior to Dropout | 3.1 [1 to 12] | 2.9 [1 to 12]

2. Primary Outcome: PTSD Checklist-Military (PCL-M)
Description: PTSD Checklist-Military (PCL-M): The PCL is a 17 Item Self Report Measure of PTSD Symptoms Based on the DSM-IV Criteria. The PCL uses a 5-point Likert scale response format ranging from not at all to frequently. The instrument is highly correlated with the Clinician Administered PTSD Scale (r = .93), has good diagnostic efficiency (> .70), and robust psychometrics with a variety of trauma populations (Blanchard, 1996), including combat veterans (Magruder, Frueh, et al, 2005). Total scores on the PCL range from 17 to 85, with lower scores indicating less symptom severity.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person
Number analyzed (Participants) | 64 | 68
score on a scale
  Average PCL Score at Baseline | 64 [17.0 to 85.0] | 61.8 [17.0 to 85.0]
  Average PCL Score at 1 week Post Tx | 48.4 [17.0 to 85.0] | 44.9 [17.0 to 85.0]
  Average PCL Score at 3 months Post Tx | 49.2 [17.0 to 85.0] | 46.5 [17.0 to 85.0]
  Average PCL Score at 6 months Post Tx | 51.7 [17.0 to 85.0] | 48.0 [17.0 to 85.0]

3. Primary Outcome: Beck Depression Inventory-II (BDI-II)
Description: Beck Depression Inventory-II (BDI-II): (BDI; Beck et al., 1961): The BDI-II is a 21-item self-report scale, is among the most widely used instruments to measure depression. Beck and Steer (1984) demonstrated that the BDI-I has high internal consistency (α = .86 - .91). Lower scores indicate less symptom severity, and higher scores indicate more severe depressive symptoms. Raw scores of 0-13 indicates minimal depression; 14-19 indicates mild depression; 20-28 indicates moderate depression; 29-63 indicates severe depression. The lowest possible score on this measure is 0, and the highest possible score is 63.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person
Number analyzed (Participants) | 64 | 68
score on a scale
  Average BDI Score at Baseline | 28.0 [0.0 to 63.0] | 27.4 [0.0 to 63.0]
  Average BDI Score at 1 week Post Tx | 21.7 [0.0 to 63.0] | 19.6 [0.0 to 63.0]
  Average BDI Score at 3 months Post Tx | 18.3 [0.0 to 63.0] | 17.6 [0.0 to 63.0]
  Average BDI Score at 6 months Post Tx | 21.6 [0.0 to 63.0] | 18.4 [0.0 to 63.0]

4. Secondary Outcome: Clinician Administered PTSD Scale for DSM-IV (CAPS IV)
Description: The Clinician Administered PTSD Scale (CAPS) is a structured interview designed to make a categorical PTSD diagnosis, as well as to provide a measure of PTSD symptom severity. The structure corresponds to the DSM-IV criteria for PTSD diagnoses, with B, C, and D symptoms rated for both frequency and intensity; these two scores (frequency + intensity) are summed to provide severity ratings. Additional questions assess Criteria A, E, and F. It is recommended that the "1, 2" rule be used to determine whether a symptom meets criteria; that is, a frequency score of at least 1 (scale 0 = "none of the time" to 4 = "most or all of the time") and an intensity score of at least 2 (scale 0 = "none" to 4 = "extreme") is required for a particular symptom to meet criteria. Total scores from B, C and D range from 0 to 136, with lower scores indicating better outcomes, and higher scores indicating worse outcomes.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person
Number analyzed (Participants) | 64 | 68
scores on a scale
  Mean CAPS Score at Baseline | 68.4 [65.5 to 71.3] | 68.2 [64.7 to 71.6]
  Mean CAPS Score at 1 Week Post | 41.9 [34.8 to 49.2] | 41.1 [33.0 to 48.2]
  Mean CAPS Score at 3 Month Post | 41.0 [32.3 to 49.7] | 38.7 [31.8 to 45.7]
  Mean CAPS Score at 6 Month Post | 46.8 [40.0 to 53.7] | 41.0 [35.0 to 47.1]

5. Secondary Outcome: Deployment Risk and Resiliency Inventory (DRRI)
Description: The DRRI is collection of self-report measures assessing 14 key deployment-related risk and resilience factors with demonstrated implications for veterans' long-term health. With the nature of military deployment changing, with a larger proportion of women, National Guard and Reserves being deployed for more contemporary conflicts, the DRRI was developed to provide a more comprehensive assessment of the current combat-related experiences. The DRRI is made up of multiple scales to represent different constructs. Responses are either dichotomous (0=No, 1=Yes), polytomous (0=No, 1=Not Sure, 2=Yes), or recorded on a 4, 5 or 6 point Likert scales. Scores for each section are summed are contain scoring ranges. Higher scores are indicative of worse outcomes.
Time Frame: Week 0
Population: The outcome data for this measure is not available because there was not enough sufficient responses to generate analyses.
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Health Related Functioning: Medical Outcome Study (MOS) Short Study Forms-36 Health Survey (SF 36)
Description: The MOS SF-36 is an indicator of overall health status. It consists of eight scaled scores, which are the weighted sums of the questions in their section. Each of the eight summed scores is linearly transformed onto a scale from 0 (negative health) to 100 (positive health) to provide a score for each subscale. Therefore, lower scores indicate more disability while higher scores indicate less disability. Each subscale can be used independently. Sections of the SF-36 include: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person
Number analyzed (Participants) | 64 | 68
percentage of participants
  % reported very good/excellent health at Baseline | 18.60 | 10.90
  % reported very good/excellent health: 1 week F/U | 17.90 | 19.00
  % reported very good/excellent health: 3 mo. F/U | 15.00 | 12.90
  % reported very good/excellent health: 6 mo. F/U | 18.90 | 22.00

7. Secondary Outcome: Charleston Psychiatric Outpatient Satisfaction Scale (CPOSS-VA)
Description: The CPOSS is a 16-item measure, with a Likert scale response format, based on a general measure of patient satisfaction. Extant data demonstrate that the measure has excellent reliability (alpha = 0.96) and good convergent validity with relevant anchor items ("would you recommend this treatment to a friend or family member?"). Items are scored using a 5 point Likert scale (5=excellent; 4=very good; 3=good; 2=fair; 1=poor). The scale is scored by summing the scores of all individual items. The possible range is 16 to 80, with higher scores indicating higher satisfaction.
Time Frame: 14 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person
Number analyzed (Participants) | 64 | 68
score on a scale | 65.6 [59.6 to 69.3] | 65.5 [62.3 to 68.7]

8. Secondary Outcome: Treatment Credibility
Description: This measures assesses for differences in outcome expectancy. The Treatment Credibility Scale (as used in this study) contains 4 questions. Each question is scored individually via 10-point Likert scales. Questions asses how logical treatment seems, how confident participants are about treatment, and expectations of success and is administered at treatment session 4. Scores on treatment logicality, confidence and predicted success on each question range from 1 (not at all) to 10 (very logical), with mid-range scores indicating moderate logicality, confidence and predicted success.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person
Number analyzed (Participants) | 64 | 68
scores on a scale | 4.4 [4.1 to 4.8] | 4.5 [4.3 to 4.7]

9. Secondary Outcome: Service Delivery Perceptions Questionnaire
Description: This measure is used to assess Veterans' perceptions about variables specifically related to this mode of service delivery (e.g., the quality of communication, ease of use, and willingness to use treatment via videoconferencing in the future). There are 8 questions (1 question was not assessed due to asking about group participation which is irrelevant to the current study). All questions are answered via a 5 point Likert scale, with 1 indicating poor perceptions and 5 indicating excellent perceptions. Scores range from 7-35, with higher scores indicating more positive outcomes.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person
Number analyzed (Participants) | 64 | 68
units on a scale | 4.6 [4.4 to 4.9] | 4.7 [4.5 to 4.8]

10. Secondary Outcome: Structured Clinical Interview for DSM-IV (SCID-I)
Description: The Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I) is a semistructured interview to determine whether an individual meets criteria for any Axis I disorder in the Diagnostic and Statistical Manual of Mental Disorders (version IV). The SCID is broken down into separate modules corresponding to categories of diagnoses, and uses skip logic to allow the interviewer to skip questions or modules if certain diagnostic criteria are indicated. Most sections begin with an entry question that would allow the interviewer to "skip" the associated questions if not met. For all diagnoses symptoms are coded as present, subthreshold, or absent. It assesses for both current and lifetime diagnoses and prompts the interviewer to document age of illness onset and to rate current illness severity (Glasofer et al., 2015).
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person
Number analyzed (Participants) | 64 | 68
percentage of participants
  Base SCID % Depression DX | 75.6 | 86.5
  Post SCID % Depression DX | 66.7 | 52.9
  Month 3 SCID % Depression DX | 58.3 | 40.0
  Month 6 SCID % Depression DX | 62.5 | 42.1
  Base SCID % Panic DX | 30.0 | 33.0
  Post SCID % Panic DX | 50 | 28
  Month 3 SCID % Panic DX | 40 | 20
  Month 6 SCID % Panic DX | 38.5 | 53.8

11. Secondary Outcome: Prior Experience With Computer and Audiovisual Technology
Description: The Prior Experience With Technology questionnaire is an 8-item short measure to learn more about participants' prior experiences and comfort level with computers and audiovisual technology. For 8 different technological devices, the measure asks if the participant has the device in his/her home (i.e. Is there a telephone in your home)? Subsequent questions determine whether the patient is comfortable using that device or, if he/she does not own one, if he/she would be willing to learn to use one. Devices assessed include telephone, television, stereo, video player (e.g. VCR, DVD), computer, internet, e-mail, and audiovisual conferencing technology. These data may help identify whether these variables are associated with clinical outcome.
Time Frame: Week 0
Population: as for outcome 5
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: There were 150 participants enrolled in the study, and 132 completed at least one session and were thus analyzed (see participant flow and baseline characteristics sections). We are reporting adverse event statistics on the basis of total enrollment.
Arm/Group | Arm 1: PE Via Telemedicine | Arm 2: PE in Person
Serious Adverse Events (participants affected / at risk) | 0/74 | 1/76
Other Adverse Events (participants affected / at risk) | 0/74 | 0/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: PE Via Telemedicine (N=74) | Arm 2: PE in Person (N=76)
Death (Psychiatric disorders) | 0 (0) | 1 (1) — Participant completed Prolonged Exposure treatment on 6/23/14. On 10/1/14 study staff were notified by VA clinicians that participant committed suicide on 9/30/14. Event was determined to be unexpected and unrelated to study.

LIMITATIONS AND CAVEATS:
1. The study lacked a third group of participants receiving an alternative intervention to compare PE-HBT with a standard control-group.
2. The achieved effect sizes were less than those typically evident in PE treatment outcome studies

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No